CLINICAL TRIAL: NCT05663424
Title: Comparative Efficacy of Different Time Interval Between rTMS and Rehabilitation Program for Motor Recovery in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 111-080-F
Record Dates: First submitted 2022-12-09; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Stroke
Keywords: rTMS; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- immediate rehabilitation group (Experimental): rTMS plus immediate rehabilitation programs
  Interventions: Other: rTMS-PTi
- delayed rehabilitation group (Experimental): rTMS plus delayed rehabilitation programs
  Interventions: Other: rTMS-PTd
- sham rTMS group (Sham Comparator): sham rTMS + rehabilitation programs
  Interventions: Other: rTMSs-PT

INTERVENTIONS:
Other: rTMS-PTi — 10 daily sessions of rTMS (1Hz, 1200 short, for totally 20 minutes) plus immediate rehabilitation programs
  Arms: immediate rehabilitation group
Other: rTMS-PTd — 10 daily sessions of rTMS (1Hz, 1200 short, for totally 20 minutes) plus delayed rehabilitation programs (>2hr)
  Arms: delayed rehabilitation group
Other: rTMSs-PT — 10 daily sessions of sham rTMS (to vertex) plus rehabilitation programs
  Arms: sham rTMS group

SUMMARY:
Comparative Efficacy of Different Time Interval between rTMS and Rehabilitation Program for Motor Recovery in Stroke Patients

DETAILED DESCRIPTION:
Stroke is one of the main causes of death and disability in Taiwan. The M1 excitability of the affected hemisphere decreases, while that of the unaffected hemisphere increases, leading to further interhemispheric inhibition. Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive neuromodulation technology. High and low frequencies of rTMS could modulate the excitability of the cerebral cortex. Through regulating the excitability of bilateral hemispheres, rTMS could facilitate motor recovery in stroke patients. Previous study had been demonstrated that priming rehabilitation program with low frequent rTMS would lead to better motor recovery in the chronic stroke patients. However, the optimal time interval between the rTMS and the rehabilitation program had not been investigated. Thus, this study will utilize low frequent rTMS, targeting the intact hemisphere, to investigate the clinical effects and motor cortex excitability under different time intervals between the rTMS and the rehabilitation program.

This study is designed as a randomized controlled trial. We plan to recruit 45 subacute stroke patients with hemiplegia. The patients are randomly assigned to three groups. In the Group 1, the patients receive contralateral 1 Hz rTMS stimulation and subsequent rehabilitation program. In the Group 2, the patients receive contralateral 1 Hz rTMS, but the rehabilitation will be delayed at least two hours after the rTMS stimulation. The control group receive sham rTMS and subsequent rehabilitation program. The treatment schedule for all groups will be five times per week for a two-week course, which means a total of ten sessions. The primary outcome is upper limb Fugl-Meyer Assessment. The secondary outcomes included Medical Research Council (MRC) scale, Barthel Scale, Modified Rankin Scale (MRS), cortical excitability assessment (including bilateral maximum MEP amplitude, MEP latency, and bilateral resting motor threshold). Follow-up time points are before rTMS and at 1st, 4th, 12th weeks after the end of the treatments.

ELIGIBILITY:
Inclusion criteria

1. >=20 years old, unilateral stroke diagnosed by CT or MRI
2. Post-stroke 1 week to 6 months
3. Medical Research Council Scale for Muscle Strength in upper limb ≤ 3
4. No history of previous stroke, seizure, dementia, parkinsonism or other neurodegenerative disease
5. stable medical condition and vital signs

Exclusion criteria

1. Previous stroke, traumatic brain injury, brain tumor
2. With central nervous system disease (spinal cord injury, Parkinson's disease)
3. Any contraindication to rTMS (seizure, alcoholism, metal implant, pacemaker, Pregnancy...)
4. Patients unable to cooperate the treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (FMA) | 12 weeks
  Fugl-Meyer Assessment (FMA) of upper limb

SECONDARY OUTCOMES:
Medical Research Council (MRC) scale | 12 weeks
  Medical Research Council (MRC) scale
Grip strength | 12 weeks
  Grip strength (Kg)
Barthel Index | 12 weeks
  Barthel Index
Modified Rankin Scale | 12 weeks
  Modified Rankin Scale
maximal motor evoked potential amplitude | 12 weeks
  maximal motor evoked potential amplitude of lesion site (mV)
motor evoked potential latency | 12 weeks
  motor evoked potential latency of lesion site (ms)
resting motor threshold | 12 weeks
  bilateral resting motor threshold (mV)

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Hao Cheng, MD, Principal Investigator — The Department of Physical Medicine and Rehabilitation, National Taiwan University Hospital Hsin-Chu Branch
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch, Hsinchu, Taiwan